CLINICAL TRIAL: NCT04866199
Title: Peri-Operative Metabolic & Mitochondrial Phenotype Study: Prediction From Three Preoperative Assessments
Brief Title: POM-MP: PeriOp Metabolic & Mitochondrial Phenotype
Acronym: POM-MP
Status: Withdrawn | Type: Observational
Why Stopped: Key investigator left institution
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00108362
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Surgical Complications From Surgery; Surgical Complications From Bladder Surgery; Surgical Complications From Bowel Surgery
Keywords: Surgery; Complication; Preoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples 30 mL taken at Baseline (preop), Postop Days 0, 1, 3 & 5 and up to Postop Day 30. Total 180 mL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High-risk colon or bladder surgical patients: Patients who are diagnosed with colon or bladder cancer requiring surgical resection.

SUMMARY:
Patients scheduled for bladder or bowel resection will receive assessments at three time points:

1. Preoperatively up to 30 days prior to scheduled surgery
2. Postoperatively in hospital up to 5 days
3. Postoperatively up to 30 days following scheduled surgery

At all time points the subjects will have blood samples drawn for mitochonrial function analysis and a muscle ultrasound (MuscleSound) performed. In addition, a cardiopulmonary exercise test (CPET or 'VO2 max') will be performed at the 30 day pre/post evaluation time points.

DETAILED DESCRIPTION:
Cardiorespiratory fitness (CRF) is a measure of the efficiency to use oxygen. One method used to measure CRF is the cardiopulmonary exercise test (CPET), otherwise known as 'VO2 max'. Previous studies have shown that individuals assessed with CPET-derived parameters, such as VO2 max or anaerobic threshold (AT), below specific thresholds are at greater risk of post-operative complications, which can occur in up to 40% of surgical patients.

This study wants to determine if other methods of fitness or well-being, such as mitochondrial oxygen consumption and muscle ultrasound to determine muscle characteristics, can be combined with CPET assessment to improve the ability to identify surgical patients who develop postoperative complications, as measured by the validated tool, POMS.

The objective of the study is to create a method to identify the metabolic and mitochondrial phenotype of the perioperative patient, termed the POM-MP.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged >18 undergoing bladder or bowel resection
* Able to speak English
* Ambulatory (assistive devices OK)
* Able to consent
* Willing to perform Cardiopulmonary Exercise Testing

Exclusion Criteria:

* Unable to perform CPET
* Pregnant
* Prisoner
* Patients with diagnosed Dementia
* Unable to ambulate independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients identified in surgical clinic as candidates for bladder or bowel resection.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with post-operative complications as measured by Postoperative Morbidity Survey (POMS) | Up to 30 days post-op
  Nine-domain tool used to assess the presence (or absence) of clinically significant changes using specified criteria. Confirmation of yes in any domain represents post-operative morbidity.
Change in the highest oxygen consumption (VO2 peak) as measured by wearable face mask | Baseline (preop) and Post-op (up to 30 days)
  Measured in milliliters of oxygen per min
Change in MuscleSound %iMAT as measured by portable ultrasound | Baseline (preop), postop Days 0, 1, 3 & 5, and Post-op (up to 30 days)
  The parameter is derived using a proprietary algorithm applied to the ultrasound image to estimate the amount of intramuscular adipose tissue, presented as percentage
Change in mitochondrial oxygen consumption as measured by blood analysis | Baseline (preop), postop Days 0, 1, 3 & 5, and Post-op (up to 30 days)
  The change between baseline and maximal oxygen consumption when maximum induced by additon of chemicals in vivo

CONTACTS AND LOCATIONS:
Overall Officials: David B MacLeod, FRCA, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No